CLINICAL TRIAL: NCT01007123
Title: A Phase IIb, Double-blind, Randomised, Placebo-controlled, Multi-centre, Dose-finding Efficacy and Safety Study of a Range of Doses of Elobixibat in Patients With Chronic Idiopathic Constipation
Brief Title: Study of Elobixibat (A3309) in Patients With Chronic Idiopathic Constipation
Acronym: ACCESS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Albireo (Industry)
Responsible Party: Sponsor
Organization: AlbireoPharma (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A3309-002
Record Dates: First submitted 2009-11-02; First posted 2009-11-03 (Estimated); Results first posted 2017-03-22 (Actual); Last update posted 2017-03-22 (Actual); Status verified 2017-02

CONDITIONS: Constipation; Chronic Constipation
Keywords: Chronic idiopathic constipation; A3309
MeSH Terms: conditions — Constipation | interventions — elobixibat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- A3309 low dose (Experimental): Administered once daily for the duration of the study
  Interventions: Drug: A3309
- A3309 intermediate dose (Experimental): Administered once daily for the duration of the study.
  Interventions: Drug: A3309
- A3309 high dose (Experimental): Administered once daily for the duration of the study
  Interventions: Drug: A3309
- Placebo (Placebo Comparator): Administered once daily for the duration of the study
  Interventions: Drug: A3309

INTERVENTIONS:
Drug: A3309 — A3309 in three different dosage levels or placebo once daily for the duration of the study

SUMMARY:
The purpose of this trial is to determine the efficacy and safety of A3309 administered to patients with chronic idiopathic constipation.

ELIGIBILITY:
Inclusion Criteria:

* Patient meets protocol specified criteria for constipation
* Patient has successfully completed study requirements with no clinically relevant findings for physical exam, ECG, laboratory tests and colonoscopy as applicable

Exclusion Criteria:

* Medical history or medical condition that would not make the patient a good candidate for the study or limit the patient´s ability to complete the study
* Patient reports loose stools
* Patient has IBS with pain/discomfort as predominant symptom
* Patient needs medications prohibited as specified in the protocol

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2009-11; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hans Graffner, MD, Study Chair — Albireo
Locations (43):
- United States (43):
  - Albireo Investigative Site, Huntsville, Alabama
  - Albireo Investigative Site, Chandler, Arizona
  - Albireo Investigative Site, Phoenix, Arizona
  - Albireo Investigative Site, Anaheim, California
  - Albireo Investigative Site, Encinitas, California
  - Albireo Investigative Site, San Diego, California
  - Albireo Investigative Site, Colorado Springs, Colorado
  - Albireo Investigative Site, Boynton Beach, Florida
  - Albireo Investigative Site, Inverness, Florida
  - Albireo Investigative Site, Peoria, Illinois
  - Albireo Investigative Site, Clive, Iowa
  - Albireo Investigative Site, Davenport, Iowa
  - Albireo Investigative Site, Mission, Kansas
  - Albireo Investigative Site, Overland Park, Kansas
  - Albireo Investigative Site, Monroe, Louisiana
  - Albireo Investigative Site, Shreveport, Louisiana
  - Albireo Investigative Site, Annapolis, Maryland
  - Albireo Investigative Site, Baltimore, Maryland
  - Albireo Investigative Site, Hollywood, Maryland
  - Albireo Investigative Site, Chesterfield, Michigan
  - Albireo Investigative Site, Henderson, Nevada
  - Albireo Investigative Site, Marlton, New Jersey
  - Albireo Investigative Site, Albuquerque, New Mexico
  - Albireo Investigative Site, Great Neck, New York
  - Albireo Investigative Site, Charlotte, North Carolina
  - Albireo Investigative Site, Greensboro, North Carolina
  - Albireo Investigative Site, Harrisburg, North Carolina
  - Albireo Investigative Site, Statesville, North Carolina
  - Albireo Investigative Site, Winston-Salem, North Carolina
  - Albireo Investigative Site, Cincinnati, Ohio
  - Albireo Investigative Site, Dayton, Ohio
  - Albireo Investigative Site, Oklahoma City, Oklahoma
  - Albireo Investigative Site, Levittown, Pennsylvania
  - Albireo Investigative Site, Anderson, South Carolina
  - Albireo Investigative Site, Chattanooga, Tennessee
  - Albireo Investigative Site, Kingsport, Tennessee
  - Albireo Investigative Site, El Paso, Texas
  - Albireo Investigative Site, Longview, Texas
  - Albireo Investigative Site, San Antonio, Texas
  - Albireo Investigative Site, Ogden, Utah
  - Albireo Investigative Site, Salt Lake City, Utah
  - Albireo Investigative Site, Lynchburg, Virginia
  - Albireo Investigative Site, La Crosse, Wisconsin

REFERENCES:
- [Result] Chey WD, Camilleri M, Chang L, Rikner L, Graffner H. A randomized placebo-controlled phase IIb trial of a3309, a bile acid transporter inhibitor, for chronic idiopathic constipation. Am J Gastroenterol. 2011 Oct;106(10):1803-12. doi: 10.1038/ajg.2011.162. Epub 2011 May 24. PMID 21606974

RESULTS

PARTICIPANT FLOW:
Groups:
- Elobixibat (A3309) 5 mg; Elobixibat (A3309) 10 mg; Elobixibat (A3309) 15 mg; Placebo: Administered once daily for the duration of the study
Period: Overall Study
Arm/Group | Elobixibat (A3309) 5 mg | Elobixibat (A3309) 10 mg | Elobixibat (A3309) 15 mg | Placebo
Started | 48 | 47 | 48 | 47
Completed | 42 | 41 | 37 | 41
Not Completed | 6 | 6 | 11 | 6
Not completed — Adverse Event | 3 | 4 | 7 | 1
Not completed — Lack of Efficacy | 1 | 0 | 1 | 4
Not completed — Protocol Violation | 1 | 1 | 2 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Elobixibat (A3309) 5 mg | Elobixibat (A3309) 10 mg | Elobixibat (A3309) 15 mg | Placebo | Total
Number analyzed (Participants) | 48 | 47 | 48 | 47 | 190
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 44 | 46 | 43 | 41 | 174
  >=65 years | 4 | 1 | 5 | 6 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (13) | 48 (11) | 46 (13) | 50 (13) | 48 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 45 | 43 | 39 | 170
  Male | 5 | 2 | 5 | 8 | 20
Region of Enrollment [Number; unit: participants]
  United States | 48 | 47 | 48 | 47 | 190

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Frequency of Spontaneous Bowel Movements
Description: Primary ep W 1
Time Frame: Baseline, weekly, up to 8 weeks
Population: ITT population
Measure: Least Squares Mean (Standard Error); unit: Number of SBMs
Arm/Group | Elobixibat (A3309) 5 mg | Elobixibat (A3309) 10 mg | Elobixibat (A3309) 15 mg | Placebo
Number analyzed (Participants) | 46 | 43 | 44 | 46
Number of SBMs | 2.5 (0.7) | 4.0 (0.7) | 5.4 (0.71) | 1.7 (0.7)
Statistical Analysis 1: Comparison: Elobixibat (A3309) 5 mg vs Placebo; Test type: Superiority or Other; p < 0.2, ANCOVA
Statistical Analysis 2: Comparison: Elobixibat (A3309) 10 mg vs Placebo; Test type: Superiority or Other; p = 0.002, ANCOVA
Statistical Analysis 3: Comparison: Elobixibat (A3309) 15 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA

2. Secondary Outcome: Responder Analyses for Complete Spontaneous Bowel Movements (CSBMs)
Description: A CSBM responder is defined as per FDA draft guidance for IBS-C:
  An increase of one or more of CSBMs per week over baseline for at least 4 out of the 8 weeks of treatment
Time Frame: Baseline, weekly and up to 8 weeks
Population: ITT population
Measure: Number; unit: participants
Arm/Group | Elobixibat (A3309) 5 mg | Elobixibat (A3309) 10 mg | Elobixibat (A3309) 15 mg | Placebo
Number analyzed (Participants) | 43 | 42 | 40 | 42
participants | 25 | 27 | 30 | 14
Statistical Analysis 1: Comparison: Elobixibat (A3309) 5 mg; Test type: Superiority or Other; p = 0.03, Fisher Exact
Statistical Analysis 2: Comparison: Elobixibat (A3309) 10 mg vs Placebo; Test type: Superiority or Other; p = 0.008, Fisher Exact
Statistical Analysis 3: Comparison: Elobixibat (A3309) 15 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Fisher Exact

3. Secondary Outcome: Time to First Bowel Movement
Time Frame: First week
Population: ITT population
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Elobixibat (A3309) 5 mg | Elobixibat (A3309) 10 mg | Elobixibat (A3309) 15 mg | Placebo
Number analyzed (Participants) | 40 | 39 | 40 | 40
hours | 23 [17 to 29] | 12 [7 to 23] | 7 [5 to 20] | 27 [20 to 44]
Statistical Analysis 1: Comparison: Elobixibat (A3309) 5 mg vs Placebo; Test type: Superiority or Other; p = 0.06, Fisher Exact
Statistical Analysis 2: Comparison: Elobixibat (A3309) 10 mg vs Placebo; Test type: Superiority or Other; p = 0.03, Fisher Exact
Statistical Analysis 3: Comparison: Elobixibat (A3309) 15 mg vs Placebo; Test type: Superiority or Other; p = 0.04, Fisher Exact

4. Secondary Outcome: Stool Consistency Change From Baseline
Description: Bristol Stool Form Scale. Min value:1. Max value: 7. Higher value indicates more liquid shape than normal, lower indicates constipated state.
Time Frame: Baseline, weekly and up to 8 weeks
Population: ITT population
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale (1-7)
Arm/Group | Elobixibat (A3309) 5 mg | Elobixibat (A3309) 10 mg | Elobixibat (A3309) 15 mg | Placebo
Number analyzed (Participants) | 48 | 47 | 48 | 47
units on a scale (1-7) | 0.91 (0.99) | 1.52 (1.2) | 1.91 (1.3) | 0.66 (1.0)
Statistical Analysis 1: Comparison: Elobixibat (A3309) 5 mg vs Placebo; Test type: Superiority or Other; p = 0.44, ANCOVA
Statistical Analysis 2: Comparison: Elobixibat (A3309) 10 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 3: Comparison: Elobixibat (A3309) 15 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA

5. Secondary Outcome: LDL/HDL Ratio
Description: Ratio of plasma LDL cholesterol and HDL cholesterol Difference from baseline, placebo-adjusted
Time Frame: Baseline and 8 weeks of treatment
Population: ITT population
Measure: Least Squares Mean (Standard Error); unit: Ratio
Groups:
- Eobixibat (A3309) 10 mg; Elobixibat (A3309) 15 mg: Administered once daily for the duration of the study.
Arm/Group | Elobixibat (A3309) 5 mg | Eobixibat (A3309) 10 mg | Elobixibat (A3309) 15 mg
Number analyzed (Participants) | 48 | 46 | 48
Ratio | -0.10 (0.08) | -0.27 (0.09) | -0.21 (0.1)
Statistical Analysis 1: Comparison: Eobixibat (A3309) 10 mg; Comparison vs placebo; Test type: Superiority or Other; p = 0.01, ANCOVA
Statistical Analysis 2: Comparison: Elobixibat (A3309) 15 mg; Comparison vs placebo; Test type: Superiority or Other; p < 0.05, ANCOVA

6. Secondary Outcome: Straining Change From Baseline
Description: Daily assessment of straining. Min value: 1. Max value: 5. Higher value indicates more straining.
Time Frame: Baseline and during 8 weeks of treatment
Population: ITT population
Measure: Least Squares Mean (Standard Error); unit: units on a scale (1-5)
Arm/Group | Elobixibat (A3309) 5 mg | Elobixibat (A3309) 10 mg | Elobixibat (A3309) 15 mg | Placebo
Number analyzed (Participants) | 48 | 46 | 48 | 47
units on a scale (1-5) | -0.84 (0.1) | -1.13 (0.1) | -1.15 (0.1) | -0.64 (0.1)
Statistical Analysis 1: Comparison: Elobixibat (A3309) 5 mg vs Placebo; Test type: Superiority or Other; p = 0.17, ANCOVA
Statistical Analysis 2: Comparison: Elobixibat (A3309) 10 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 3: Comparison: Elobixibat (A3309) 15 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA

ADVERSE EVENTS:
Time Frame: From randomization to end of follow-up 14 days after end of treatment
Arm/Group | Elobixibat (A3309) 5 mg | Elobixibat (A3309) 10 mg | Elobixibat (A3309) 15 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 1/48 | 1/47 | 0/48 | 1/47
Other Adverse Events (participants affected / at risk) | 5/48 | 5/47 | 13/48 | 3/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Elobixibat (A3309) 5 mg (N=48) | Elobixibat (A3309) 10 mg (N=47) | Elobixibat (A3309) 15 mg (N=48) | Placebo (N=47)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Cancer diagnosed 5 days after treatment start Not considered related to study drug
Bleeding colonic diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Colonoscopy verified bleeding diverticulum 14 days after end of treatment. Not considered related to study drug
Shoulder pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Not considered related to study drug
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Elobixibat (A3309) 5 mg (N=48) | Elobixibat (A3309) 10 mg (N=47) | Elobixibat (A3309) 15 mg (N=48) | Placebo (N=47)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 3 (3) | 6 (6) | 1 (46)
Abdominal pain (Gastrointestinal disorders) | 5 (5) | 5 (5) | 13 (13) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 4 (4) | 2 (2) | 3 (3) | 1 (1)
Flatulence (Gastrointestinal disorders) | 4 (4) | 3 (3) | 2 (2) | 3 (3)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less